CLINICAL TRIAL: NCT01407354
Title: Lokomat and Aquatic Therapy in Chronic Motor Incomplete Spinal Cord Injury
Brief Title: Comparison of Lokomat and Aquatic Exercise for Individuals With Chronic Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Shepherd Center, Atlanta GA (Other)
Responsible Party: Principal Investigator, Peter Gorman, Associate Professor, Neurology, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00047439; SC090147
Record Dates: First submitted 2011-07-12; First posted 2011-08-02 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injury
Keywords: robotic weight support; aquatic exercise; incomplete motor spinal cord injury; ASIA C and D
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lokomat Training (Experimental): Lokomat robotic assisted treadmill training Lokomat Treadmill Training
  Interventions: Device: Lokomat treadmill training
- Aquatic Therapy (Active Comparator): Aquatic exercise therapy
  Interventions: Other: Aquatic exercise therapy

INTERVENTIONS:
Device: Lokomat treadmill training — Lokomat treadmill training: 12 wks, 3x/wk, 45 mins@session
  Other Names: Robotic Body Weight Supported Locomotor Training
  Arms: Lokomat Training
Other: Aquatic exercise therapy — Aquatic exercise training: 12 wks, 3x/wk, 45 mins@session
  Other Names: Aquatic Therapy
  Arms: Aquatic Therapy

SUMMARY:
Many people with spinal cord injury (SCI) hold some ability to move their leg muscles, and are therefore considered to demonstrate a motor incomplete injury. After such a spinal cord injury, individuals are able to walk less both in their home and in their community. De-conditioning, or a lack of endurance and fitness also occurs. Several methods are available to try to improve walking ability and the fitness of persons with motor incomplete spinal cord injury. This study examines two of these methods. The first is the use of robotically assisted body-weight supported walking using a device called the Lokomat. The second is aquatic or pool-based exercise. The investigators are researching the impact of these two techniques on walking ability and fitness in people who experienced motor incomplete spinal cord injury for at least 12 months.

DETAILED DESCRIPTION:
This research will occur in two centers Kernan Orthopedics and Rehabilitation Hospital in Baltimore, Maryland and Shepherd Center in Atlanta, Georgia. A total of 36 volunteers over a three year period are needed. In order to qualify for this study, individuals must be 18 to 65 years old with a motor incomplete SCI. The level of injury can range from the fourth cervical level in the neck to the twelfth thoracic level in the back. Potential volunteers must be able to tolerate standing in a standing frame for at least 30 minutes. Individuals will be assessed by a physician to determine their eligibility for the study and if participating in this type of exercise would be safe. Participants must be able to understand the study requirements and sign an informed consent document.

Participants will need to commit to a total of seven months. Included in this time is: testing, then the 3 months of exercise, testing, 2 week break, then the second 3 months of exercise, and a final testing. Half of the group will start with the Lokomat training and half will start wtih aquatic exercise. Each group will then switch to the other exercise condition. Exercise sessions will occur three times per week and last approximately 45-55 minutes. A physical therapist will provide personal direction for each of the exercise groups. Walking ability and cardiovascular fitness, as well as muscle strength will be assessed before starting exercise, at the three-month point and then at the six month point.

It is hoped that that this type of exercise therapy will help individuals with motor incomplete spinal injury both walk better and experience better heart-lung fitness and endurance. The risks associated with this type of study are similar to any type of cardiovascular exercise. In addition, individuals with spinal cord injury may present with some medical conditions, there may be other risks of the study. The physicians and therapists involved in the research will discuss these risks in detail with the individuals who enroll.

This type of research is important to better understand how best to prescribe exercise treatments to people with spinal injury. This is especially true with regards to aquatic therapy, since there is very little scientific data on its effect in this group of individuals. The rigorous assessment of aquatic exercise, which is already available in many communities, may expand the fitness opportunities for individuals with incomplete spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Level of injury between C4 and T12 based on ASIA classification
* Chronic (greater than 12 months) spinal injury
* Completion of all conventional inpatient rehabilitation therapy
* Motor incomplete spinal cord injury (AIS C or D)
* Competency to provide informed consent
* Ability to tolerate a standing frame for at least 30 minutes

Exclusion Criteria:

* Currently performing aquatic therapy or Lokomat training as part of clinical care
* Complete or concurrent lower motor neuron injury as defined by the absence of reflexes bilaterally at the knees and the ankles
* Uncontrolled seizures
* Skin opening greater than 2 cm in diameter
* Alcohol consumption > 3 oz liquor, or 3 x 4oz of wine, or 36 oz of beer per day
* Cardiac history of (a) unstable angina, (b) recent (< 3 months) myocardial infarction, (c) congestive heart failure (NYHA category II), or (d) hemodynamically significant valvular dysfunction
* Medical history of (a) recent hospitalization for severe disease or surgery, (b)undiagnosed diabetics (fasting glucose > 120) or poorly controlled diabetics (those not on a stable regimen for >6 months) unable to be controlled with medical treatment, (c) significant orthopedic or chronic pain conditions limiting exercise, (d) active neoplastic disease, (e) pulmonary or renal disease, and (f) presence of any serious medical condition with a prognosis for death or dependency in the next 2 months
* History of long bone fracture in the legs
* Frequent bouts of autonomic dysreflexia (as determined by the principal investigator)
* Any other medical co-morbidities that based on the judgment of the local principal investigator would preclude safe participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Geigle, PT, PhD, Principal Investigator — University of Maryland Rehabilitation and Orthopaedic Institute; Peter H Gorman, MD, FAAN, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - Shepherd Center, Virginia C. Crawford Research Institute, Atlanta, Georgia
  - University of Maryland Rehabilitation & Orthopaedic Institute (formerly known as Kernan Hospital), Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorman PH, Scott W, VanHiel L, Tansey KE, Sweatman WM, Geigle PR. Comparison of peak oxygen consumption response to aquatic and robotic therapy in individuals with chronic motor incomplete spinal cord injury: a randomized controlled trial. Spinal Cord. 2019 Jun;57(6):471-481. doi: 10.1038/s41393-019-0239-7. Epub 2019 Jan 18. PMID 30659286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinicaltrial.gov, facility IRB approved SCI database, medical community all helped recruit for this study
Pre-assignment Details: Randomized Controlled Trial (which arm to initiate study) cross over design with no wash out period between arms. Adjusted statistically for change in each arm and arm participation order.
Groups:
- Lokomat First Then Aquatic Exercise: Lokomat robotic assisted treadmill training Lokomat Treadmill Training
  Lokomat treadmill training: Lokomat treadmill training: 12 wks, 3x/wk, 45 mins@session, participants received aquatic exercise after lokomat
- Aquatic Therapy First Then Lokomat Intervention: Aquatic exercise therapy
  Aquatic exercise therapy: Aquatic exercise training: 12 wks, 3x/wk, 45 mins@session, participants received lokomat intervention after aquatic exercise
Period: First Intervention
Arm/Group | Lokomat First Then Aquatic Exercise | Aquatic Therapy First Then Lokomat Intervention
Started | 20 | 17
Completed | 18 | 15
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Second Intervention
Arm/Group | Lokomat First Then Aquatic Exercise | Aquatic Therapy First Then Lokomat Intervention
Started | 18 | 15
Completed | 18 | 13
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Baseline data reflects all participants who received both aquatic exercise and lokomat training during the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 11
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Demonstrating 10% Change: Arm Ergometer and Lokomat Metabolic Cart VO2 Peak
Description: Peak VO2 via Arm Ergometer and Lokomat with metabolic cart
Time Frame: 7 months
Measure: Number; unit: participants
Arm/Group | Lokomat Training | Aquatic Therapy
Number analyzed (Participants) | 31 | 33
participants
  Number of participants with 10% changePeak VO2 Arm | 17 | 13
  number participants with 10% changPeak VO2 lokomat | 17 | 12

2. Secondary Outcome: Number of Movement Recorded by Activity Monitor (SAM)
Description: SAM movements not just steps were gathered one time pre, crossover and post and worn on ankle for 5 days; percent change for each intervention
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: number of movements
Groups:
- Lokomat: Lokomat robotic assisted treadmill training Lokomat Treadmill Training
  Lokomat treadmill training: Lokomat treadmill training: 12 wks, 3x/wk, 45 mins@session,
Arm/Group | Lokomat | Aquatic Therapy
Number analyzed (Participants) | 31 | 33
number of movements | 61141 (1823) | 82692 (1785)
Statistical Analysis 1: Comparison: Lokomat vs Aquatic Therapy; Test type: Superiority or Other; p = 0.05, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Lokomat vs Aquatic Therapy; Test type: Superiority or Other; p = 0.024, Wilcoxon (Mann-Whitney); threshold p value for statistical significance=0.05

ADVERSE EVENTS:
Arm/Group | Lokomat Training | Aquatic Therapy
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 2/37 | 1/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lokomat Training (N=37) | Aquatic Therapy (N=37)
Autonomic Dysreflexia (Nervous system disorders) | 1 | 0 — inappropriate blood pressure response to exercise
parasthesia (Nervous system disorders) | 1 | 0 — pins and needles in non distribution pattern reported
medical instability (Blood and lymphatic system disorders) | 0 | 1 — unstable blood pressure unrelated to aquatic intervention. participant returned to primary care to stabilize medical condition unrelated to study......

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No